CLINICAL TRIAL: NCT05083897
Title: Effect of Hip Adductors Isometric Contraction on Knee Extensors Isokinetic Torque in Patellofemoral Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Badr University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Ramadan, teaching assistant, Badr University
Other Study IDs: yasmine zaki
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: PFPS
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 30 patients in 1 group: measuring the effect of isometric hip adduction with knee extension on the peak torque of knee extensors
  Interventions: Other: hip adduction isometric contraction

INTERVENTIONS:
Other: hip adduction isometric contraction — addition of isometric hip adduction contraction to the knee extension for measuring knee extension peak torque by the isokinetic dynamometer

SUMMARY:
the study will be done to investigate the effect of hip adduction isometric contraction on the pain level by VAS and knee extensors peak torque by using the isokinetic dynamometer in patients with unilateral patellofemoral pain syndrome

DETAILED DESCRIPTION:
the study will be done to investigate the effect of isometric hip adduction that will be measured by the hand held dynamometer (the manual muscle tester) to measure the produced adduction torque and its effect on the peak torque of knee extension by the knee extensors which will be measured by the isokinetic dynamometer in addition to measuring the pain intensity before and through the assessment by using the visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Anterior or retro-patellar knee pain from at least 2 of the following Activities: (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping (Tyler et al., 2006).
* Insidious onset of symptoms unrelated to a traumatic incident and persistent for at least 6 weeks (subacute or chronic pain).
* They will be diagnosed as a PFPS case by a physician
* The patient's age will be ranged from 18-35 years to limit the possibility that PFPS over age 35 may have been complicated by arthritic changes, and also the patients should have closed epiphyseal growth plates (Robinson and Nee, 2007).

Exclusion Criteria:

* A history of any of the following condition: meniscal or other intra articular pathologic conditions; cruciate or collateral ligament involvement.
* A history of traumatic patellar subluxation or dislocation.
* Previous surgery in the knee and hip joints.
* Any lower limb bony/congenital deformity.
* Ankle, Knee and hip joints osteoarthritis.
* A history of any conditions affects muscle strength: diabetes mellitus, rheumatoid arthritis.
* Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients suffering from unilateral patellofemoral pain syndrome
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
peak torque of knee extensors | 2 months
  the maximum rotatory force that can be generated by the knee extensor muscles measured by the isokinetic dynamometer
pain level at the patellofemoral area | 2 months
  pain will be measured around the patellofemoral area by the visual analogue scale
hip adduction peak torque | 2 months
  hip adduction maximum rotatory force measured by the hand held dynamometer

IPD SHARING:
Plan to Share IPD: Undecided
the outcomes can be used in future researches concerning this field of interest